CLINICAL TRIAL: NCT02862418
Title: Lung Imaging With Ultra-short Echo Time MRI
Brief Title: Imaging of Lungs With a New Type of Magnetic Resonance Imaging (MRI) Called UTE (Ultrashort Echo Time)
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CIN001-Lung UTE MRI
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Disease
Keywords: MRI; UTE MRI; Pulmonary
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pulmonary disease: UTE MRI
  Interventions: Other: UTE MRI
- Control: UTE MRI
  Interventions: Other: UTE MRI

INTERVENTIONS:
Other: UTE MRI — One MRI with UTE settings will be acquired.

SUMMARY:
This research study has 2 purposes:

1. To learn about new ways to use Magnetic Resonance Imaging (MRI) to take clearer pictures of the lungs. A type of MRI called Ultra Short Echo Time (UTE) will be used as well as traditional MRI.
2. To collect images and health information about lungs that have different kinds of lung diseases to compare to healthy lungs. This collection will help researchers and clinicians to better understand lung variations in health and disease.

This study will involve one MRI session that will take about 10 to 30 minutes and for some participants a breathing test that measures how well the lungs are working. This test is called spirometry.

DETAILED DESCRIPTION:
Interstitial, obstructive, and rare lung diseases are pulmonary disorders that comprise more than 300 disease entities that are poorly understood, diagnosed, and treated. X-ray computed tomography (CT) is the imaging gold standard and the current clinical practice for imaging lung structure and function of patients. Recent advances in magnetic resonance imaging (MRI) pulse sequences and hardware with ultra short echo times (UTE) have enabled MRI of lung anatomy nearly comparable to CT without the risk of ionizing radiation.

The overreaching goals of this study are:

1. to allow for technical development and validation of UTE MRI sequences as an imaging alternative to CT as well as a future diagnostic tool, and
2. to allow for preliminary UTE data generation for healthy and various disease populations. We anticipate this as being particularly important for data on children where variability is greater due to normal variations in size, age and maturity as well as distinctive differences in expression of lung diseases in pediatrics versus adult populations.

This is a prospective, controlled study for technical development and validation of UTE MRI techniques with normal and disease cohorts. This study will use the standard MRI hardware (FDA approved coils and magnet) but will be developing and refining techniques used in the MRI sequences to obtain UTE images. This refinement includes varying the MRI settings to maximize image signal, to control image contrast, and to develop the software needed to acquire more specialized images for the purpose of improved imaging of the lungs. The data will also be used to collect normative data for comparison with lung pathologies.

Subjects may enroll more than once (with separate consent). For these subjects the MRI information may be used to generate data for in-subject temporal variability in both healthy controls and disease groups.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent or Parental Permission
* Age ≥ 5 years
* Willing and able to comply with MRI instructions

Exclusion Criteria:

* History of any comorbidity reviewed at the Screening Visit that, in the opinion of the investigator, might confound the results of the study or pose an additional risk to the subject.
* Standard MRI exclusion criteria as set forth by the Cincinnati Children's Hospital Radiology Department and Imaging Research Center.
* Pregnancy

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults age 5 and older with and without diagnosed pulmonary disease.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2015-10; Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Comparison Anatomic MRI to UTE MRI | Day 1 after MRI
  UTE MR imaging sequences will be evaluated by a radiologist for image quality and, if applicable, will be compared to anatomic scans acquired with traditional MRI settings

CONTACTS AND LOCATIONS:
Overall Officials: Zackary Cleveland, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Penny New, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
MRI results may be shared with treating physicians to support clinical decisions if images are felt to have clinical significance.